CLINICAL TRIAL: NCT07091760
Title: The Effect of Su Jok Application on Pain, Anxiety and Comfort Levels After Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ayse Aydin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Leyla Ertekin Tastan
Record Dates: First submitted 2025-06-25; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Caesarean Section
Keywords: Caesarean section; Su Jok; Pain; Anxiety; Comfort; Nursing
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statistics expert, Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): A "Su Jok Therapy" training certificate was obtained by the researcher for the application of Su Jok as a nursing intervention. Due to the duration of action of the analgesics used, Su Jok application will be performed at least 4-6 hours after the surgical procedure. A personal information form will be filled out to determine the descriptive characteristics of the patients who meet the inclusion criteria before the application. Visual Analog Scale (VAS), Verbal Category Scale, Spielberg State Anxiety Scale and Postpartum Comfort Scale (PPCS) will be applied to determine the pain, anxiety and comfort levels of women before the application. Pain and anxiety levels will be determined 30 minutes after the Su Jok massage and seed application, and pain, anxiety and comfort levels will be determined 6 hours later.
  Interventions: Other: Su Jok Application
- Placebo Group (Placebo Comparator): Due to the duration of action of the analgesics used, Su Jok application will be performed at least 4-6 hours after the surgical procedure. Patients who meet the inclusion criteria will fill out a personal information form to determine their descriptive characteristics before the application. Visual Analog Scale (VAS), Verbal Category Scale, Spielberg State Anxiety Scale and Postpartum Comfort Scale (PPCS) will be applied to determine the pain, anxiety and comfort level of the woman before the application. Pain and anxiety levels will be determined 30 minutes after Su Jok massage and seed application to the area without organ reflection, and pain, anxiety and comfort levels will be determined 6 hours later.
  Interventions: Other: Placebo Application
- No Intervention : Control group (No Intervention): Due to the duration of action of the analgesics used, the patient will be interviewed at least 4-6 hours after the surgical procedure. Only routine care of the clinic will be applied to the control group. A Personal Information Form will be filled out to determine the descriptive characteristics of women who meet the inclusion criteria. Afterwards, Visual Analog Scale (VAS), Verbal Category Scale, Spielberg State Anxiety Scale and Postpartum Comfort Scale (PPCS) will be completed face to face to determine the level of pain, anxiety and comfort. Pain and anxiety levels will be determined 30 minutes after the pre-test data collection and pain, anxiety and comfort levels will be determined 6 hours later

INTERVENTIONS:
Other: Su Jok Application — The patient's hands will be preferred for the application due to the comfort and convenience of the woman after cesarean section. Su Jok therapy, massage and seed will be applied to the reflection points on the hand based on the area to be treated.
  Arms: Experimental Group
Other: Placebo Application — Placebo Intervention:
  The placebo group will be massaged and seed will be applied to an area where there is no reflection of the Su Jok organ.
  Arms: Placebo Group

SUMMARY:
Objective: To determine the effect of Su Jok application on pain, anxiety and comfort level after cesarean section. The research will be conducted as a randomized controlled experimental study with pretest-posttest control group

DETAILED DESCRIPTION:
The research population will consist of women between the ages of 18-35 who had cesarean section between September 2025 and June 2026 in the Gynecology and Obstetrics Service of Muş State Hospital. For determining the sample size of the study, in the G Power 3.1.9.4 Package Program priori power analysis was used and for repeated measures, analysis of variance was used. It was determined that the sample size required for the study to exceed 80% power at a significance level of 0.05 with a 95% confidence interval and a medium effect size was 28. Considering the possibility of the women included in the study to leave the study voluntarily and to develop complications after cesarean delivery, it is planned to take 90 people (30 intervention, 30 placebo and 30 control). Inclusion criteria: Being between 18-35 years of age, having at least primary school education, not having any health problems (such as hypertension, tuberculosis, cancer), not having hearing and vision problems, having a cesarean section with regional anesthesia, being within the first 48 hours after the operation, not having any wounds or infectious diseases in their hands, not having a diagnosis of psychiatric disease, speaking Turkish, women who voluntarily agreed to participate in the study. Exclusion criteria: Postpartum hemorrhage, incomplete completion of the application stages, complications during the application process, voluntary withdrawal of the woman from the study. Among the women who meet the criteria for participation in the study and who voluntarily agree to participate in the study, 90 people determined according to the Protocol of Power analysis will be selected by simple randomization method. Then, it was planned to include 30 women in the intervention group, 30 women in the placebo group and 30 women in the control group by randomization method. The researcher will not be blinded due to the nature of the research. Blinding will be applied to the participants and the data statistician. Participants will not know which group they are in. When the research is completed, the data of the experimental, placebo and control groups (coded with the letters A, B and C) will be analyzed by a statistician independent of the research and the findings will be reported. This research is planned to be conducted in a double-blind study design in which the participants and the statistician will be blinded. CONSORT 2010 Flow Diagram instructions will be followed in the research process. "Personal Information Form", "Visual Analog Scale (VAS)", "Verbal Category Scale", "Spielberg State Anxiety Scale" and "Postpartum Comfort Scale" will be used to collect research data. The intervention tool used in the study; Women who have had cesarean delivery who agree to participate in the study will be determined according to the inclusion criteria and will be assigned to the intervention, placebo and control groups by randomization method. The study will start by having all three groups sign an informed consent form. Following the collection of pre-test data in the individuals included in the study; Su Jok massage and seed application will be applied to the intervention group. The placebo group will receive Su Jok massage and seed application to an area without organ reflection. The control group will receive only the routine practices of the institution without any intervention. The data will be collected by the researcher between September 2025 and June 2026 by face-to-face interview in the Gynecology and Obstetrics Service of Muş State Hospital. Filling out the forms will take an average of 5-10 minutes Process steps: Intervention group: Due to the duration of action of the analgesics used, Su Jok administration will be performed at least 4-6 hours after the surgical procedure. Patients who meet the inclusion criteria will be pre-tested before the application. In the pre-test; Personal Information Form, Visual Analog Scale (VAS), Verbal Category Scale, Spielberg State Anxiety Scale and Postpartum Comfort Scale (PPCS) will be completed face to face. After the forms are filled in, Su Jok application will be performed. Visual Analog Scale (Visual Analog Scale/VAS), Verbal Category Scale, Spielberg State Anxiety Scale, and Spielberg State Anxiety Scale will be applied 30 minutes after the end of the application and Visual Analog Scale (Visual Analog Scale/VAS), Verbal Category Scale, Spielberg State Anxiety Scale, and Postpartum Comfort Scale (PANCS) will be applied 6 hours later. Placebo Group: Due to the duration of action of the analgesics used, placebo administration will be performed at least 4-6 hours after the surgical procedure. Patients who meet the inclusion criteria will be pretested before the application. In the pre-test; Personal Information Form, Visual Analog Scale (VAS), Verbal Category Scale, Spielberg State Anxiety Scale and Postpartum Comfort Scale (PPCS) will be filled by face-to-face interviews. After the forms are filled in, Su Jok will apply massage and seed application to an area without organ reflection. Visual Analog Scale (Visual Analog Scale/VAS), Verbal Category Scale, Spielberg State Anxiety Scale and Spielberg State Anxiety Scale will be applied 30 minutes after the application and Visual Comparison Scale (Visual Analog Scale/VAS), Verbal Category Scale, Spielberg State Anxiety Scale and Postpartum Comfort Scale (PANCS) will be applied 6 hours after the application. Control Group: Due to the duration of action of the analgesics used, the patient would be interviewed at least 4-6 hours after the surgical procedure. Only routine care of the clinic will be applied to the control group. The pre-test; Personal Information Form, Visual Analog Scale (VAS), Verbal Category Scale, Spielberg State Anxiety Scale and Postpartum Comfort Scale (PPCS) will be completed by face-to-face interviews for women who meet the inclusion criteria. Visual Analog Scale (VAS), Verbal Category Scale, Spielberg State Anxiety Scale and Postpartum Comfort Scale will be administered 30 minutes after the pre-test data collection and Visual Analog Scale (VAS), Verbal Category Scale, Spielberg State Anxiety Scale and Postpartum Comfort Scale will be administered 6 hours later. PSS 25 package program will be used for coding and evaluation of the data. Number, percentage, mean and standard deviation will be used to analyze the data. Normality tests of the data will be evaluated with kurtosis and skewness coefficients. Chi-Square test and independent groups t Test / Mann-Whitney U test or ANOVA / Kruskal Wallis will be used to evaluate the averages and categorical data of the scores obtained with the scales. For repeated measurements, dependent groups t Test / Wilcoxon test or ANOVA / Fridman test will be used. A significance level of p<0.05 will be accepted. The internal validity of the scales will be determined by Cronbach α coefficient. Cohen's d/eta squared value will be calculated for t-test in dependent and independent groups for the effect size of the change in scale scores. All ethical principles will be followed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-35 years of age
* Having at least primary school education
* Not having any health problems (such as hypertension, tuberculosis, cancer)
* Not having hearing and vision problem
* Having a cesarean section with regional anesthesia
* Being within the first 48 hours after the operation
* Not having any wounds or infectious diseases in their hands
* Not having a diagnosis of psychiatric disease
* Speaking Turkish, women who voluntarily agreed to participate in the study.

Exclusion Criteria:

* Postpartum hemorrhage
* Incomplete completion of the application stages
* Complications during the application process
* Voluntary withdrawal of the woman from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — giving birth by caesarean section
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | 10 months
  There are 21 questions in this form, prepared by the researchers in line with the literature
Visual Analog Scale (VAS) | 10 months
  The Visual Analog Scale is an assessment tool in which patients mark on a 10 cm ruler. The 10 cm scale, which is a numerical pain assessment scale, starts with "No pain (0)" and ends with "Intolerable pain (10)". The patient is asked to mark the place on the line that expresses pain. The distance marked by the patient is measured by taking zero as the starting distance. In this way, the patient's pain level is determined. In this study, a horizontal VAS will be used to assess pain intensity. The reason for choosing this scale in the study is that it is easy to understand and easy to use by the participants.
Verbal Category Scale | 10 months
  The scale is based on the selection of the most appropriate word to describe the patient's pain condition. The pain of the patients is evaluated with the scoring method 'No Pain 0 points, Very Mild Pain 2 points, Mild Pain 4 points, Severe Pain 6 points, Very Severe Pain 8 points, Unbearable Pain 10 points'. The patient will be asked to select the appropriate pain level. The scale is easy to apply and easy to classify.
Spielberg State Anxiety Scale | 10 months
  This scale was developed by Spielberger et al. Developed by. The adaptation of the scale to Turkish and its validity and reliability studies were carried out by Öner and Le Compte in 1983.The scale is a 4-point Likert scale consisting of the options "not at all", "somewhat", "a lot", "completely". There are 10 direct and 10 reversed statements in the scale. Positive (increasing the total anxiety score) for items 3, 4, 6, 7, 9, 12, 13, 14, 17, 18 in the scale; 1, 2, 5, 8, 10, 11, 15, 16, 19 Negative scores (reducing the total anxiety score) are obtained for the 20th items. The highest score is 80 and the lowest score is 20. A high total score indicates that the person's anxiety level is also high.Cronbach's alpha coefficient was found to be 0.79 for state anxiety. In this study, Cronbach's Alpha value was found to be 0.83.
Postpartum Comfort Scale | 10 months
  The scale developed by Karakaplan and Yıldız (2010) to determine women's comfort after cesarean delivery and vaginal delivery is Likert-type and consists of 34 items. Each item is scored between "strongly disagree" (1 point) and "strongly agree" (5 points). The lowest score that can be obtained from the scale is 34 and the highest score is 170. The scale consists of three sub-dimensions (physical, psychosocial and sociocultural). An increase in the score obtained from the scale indicates an increase in comfort. Cronbach Alpha internal consistency coefficient was calculated as 0.78.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe AYDIN, Study Director — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No